CLINICAL TRIAL: NCT01457326
Title: Early Standardized Weight Bearing Utilizing Immersion Therapy Following Periarticular Lower Extremity Fractures: Clinical and Radiographic Outcomes
Brief Title: Early Standardized Weight Bearing Utilizing Immersion Therapy Following Periarticular Lower Extremity Fractures
Status: Terminated | Type: Observational
Why Stopped: Loss to follow-up rate too high for publication and data on completed patients does not allow for a powered analysis.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Eric Kubiak, M.D., University of Utah
Other Study IDs: 34409
Record Dates: First submitted 2011-08-22; First posted 2011-10-21 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-06

CONDITIONS: Lower Extremity Periarticular Fractures
Keywords: Immersion therapy; early weight bearing physical therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Immersion Therapy- Study: 1. Patients who participate in the immersion therapy post-operative protocol and begin progressive weight bearing at 4 weeks (study)
- Control Group: 2. Patients who undergo the traditional 10-week non-weight bearing post-operative care protocol (control)

SUMMARY:
The purpose of this prospective study is evaluate the effect of a standardized early weight bearing physical therapy protocol that utilizes immersion therapy on the clinical outcomes of lower extremity periarticular fractures. The investigators null hypothesis is that the early weight bearing protocol will have the same effect as a traditional 10-week non-weight bearing protocol on clinical outcomes.

DETAILED DESCRIPTION:
Fractures of the lower extremity are common injuries that can lead to temporary or permanent disability.13 Fracture healing, regardless of treatment, is a multifactorial process that is influenced by time, biomechanics, and host biology (among other variables). The degree, timing, progression, and type of weight bearing after fractures involving the pelvis and lower extremities is an area of debate in the clinical management of a broad spectrum of orthopedic injuries.1,2,4-9,11,15 Periarticular fractures of weight bearing joints are an area of particular interest with regard to post-operative weight bearing due to the prolonged periods that patients must be non-weight bearing after surgery.

Some degree of impairment is inevitable with any traumatic injury. The majority of authors writing about post-fracture weight bearing have determined that timing and extent of weight bearing has an effect on fracture healing, while a small number of authors have published results demonstrating the opposite.14,16,19,21 In addition to potential impacts on healing rates, limited or non-weight bearing carries the added insult of loss of bone density and muscle mass.3,10,12,17,20,22

Traditionally, patients with periarticular fractures have been required to be non-weight bearing on their effected extremity for up to 12 weeks. At this institution, most patients have been required to remain non-weight bearing for 10 weeks, followed by progressively increased levels of weight bearing according to patient tolerance. One of the orthopaedic traumatologists at this institution uses immersion therapy to allow patients with periarticular fractures to begin weight bearing prior to the ten-week mark.

Immersion therapy requires that patients perform their physical therapy, with a trained therapist, in a swimming pool. The use of the pool in post-fracture care may be able to provide a structured and standardized partial weight-bearing environment that could allow for early mobilization. It also has the potential to improve clinical outcomes by mitigating at least some of the loss in bone and muscle mass during the post-operative period; thereby, potentially speeding functional recovery. Immersion therapy is currently utilized on-site at the University of Utah Orthopedic Center for a variety of diagnoses, including in post-fracture care.

There is essentially no orthopedic literature regarding immersion therapy in the management of post-fracture rehabilitation with regard to early weight bearing. Specifically, the investigators are aware of no clinical outcome studies that investigate standardized early weight bearing protocols following periarticular fractures of the lower extremity.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the patient population under study consists of both male and female adults, at least 18 years old, who are treated for periarticular fractures of the lower extremity. The periarticular fractures included in this study will be: acetabular, tibial plateau, tibial plafond fractures.

Exclusion Criteria:

* Age <18 years
* Wound complications deemed to be unsafe for immersion.
* Multiple extremity articular fractures
* Other injuries that preclude their safe participation in physical therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a prospective cohort study with a retrospective chart review. Patients who are treated by the PI, Dr. Erik Kubiak, will participate in an immersion therapy post-operative protocol. Immersion therapy post-operative protocols have been and are currently used routinely by Dr. Kubiak.
  Patients who are treated by Dr. Dan Horwitz and Dr. Thomas Higgins will undergo a traditional 10 week non-weight bearing post-operative care per their standard of procedure. In addition, patients of Dr. Kubiak who are unable to participate in immersion therapy for logistical reasons will be asked to participate in the traditional 10- week non-weight bearing post-operative care protocol. These patients will make up the control cohort.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2009-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Immersion Therapy | 10 weeks
  1. Standard ROM while in the hospital
  2. two weeks of immersion therapy, patients perform their physical therapy immersed in the pool to their neck (5-10% total body weight).
  3. weeks 6-8, patients are immersed to their mid-chest (nipple level- 15-30% total body weight).
  4. weeks 8-10, patients are progressed to physical therapy while immersed only to their waist (navel level- 50-60% total body weight).
  5. ten weeks, patients are allowed to weight bear as tolerated and begin formal dry land ambulation training under the supervision of a licensed physical therapist .
Traditional non-weightbearing | 10 weeks
  1. ROM therapy initiated in the hospital.
  2. Passive Motion therapy for 4 weeks.
  3. Formal physical therapy continued as needed

SECONDARY OUTCOMES:
Short Musculoskeletal Function Assessment | 1 year
  * Time to return to work. Assessed at each clinical visit, and by mailings if necessary.
  * Standard radiographs will be obtained from the study patients per usual at post-operative visits. Any loss of fixation will be assessed. No additional radiographs will be obtained outside of the current standard of care.
  * Adverse events will be tabulated.
  * The short Musculoskeletal Function Assessment (SMFA) will be administered at patient's 3 month, 6 month and 1 year follow-up clinic appointments and/or by mail, as necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Kubiak, MD, Principal Investigator — University of Utah Orthopedics
Locations (1):
- University of Utah Orthopedics Center, Salt Lake City, Utah, United States